CLINICAL TRIAL: NCT03269799
Title: The Effect of Vitamin C as an Adjunct in Periodontal Treatment in Uncontrolled Type 2 Diabetes Mellitus Patients
Brief Title: Vitamin C as an Adjunct in Periodontal Treatment in Type 2 Diabetes Mellitus Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Supanee Rassameemasmaung, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016/DT068
Record Dates: First submitted 2017-08-28; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus Type 2 With Hyperglycemia; Periodontitis
Keywords: uncontrolled type 2 diabetes mellitus; periodontitis; non surgical periodontal treatment; vitamin C
MeSH Terms: conditions — Periodontitis | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Active Comparator): vitamin C 500 mg oral capsule
  Interventions: Drug: Vitamin C 500 MG Oral Capsule
- control group (Placebo Comparator): placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Vitamin C 500 MG Oral Capsule — non surgical periodontal treatment+vitamin C 500 mg/day for 2 months
  Arms: test group
Other: placebo — non surgical periodontal treatment+placebo for 2 months
  Arms: control group

SUMMARY:
Periodontitis patients with uncontrolled type 2 diabetes mellitus will receive non-surgical periodontal treatment and then be supplemented with daily 500 mg vitamin C (test group) or placebo (control group) for 2 months. Clinical parameters will be retrieved at baseline, at the end of week 4 and at the end of week 8.

ELIGIBILITY:
Inclusion Criteria:

* uncontrolled type 2 diabetes mellitus
* periodontitis

Exclusion Criteria:

* complications from diabetes mellitus, e.g., renal insufficiency
* receive insulin
* diseases that interfere with wound healing, e.g., HIV
* receive one of the followings: tetracycline, acetaminophen, NSAID, warfarin, aluminum-containing antacids, barbiturates, phenobarbital, pentobarbital, secobarbital, hormone replacement therapy, chemotherapeutic drug, protease inhibitor
* receive other vitamins or antibiotics within 6 months
* smoking
* pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08-30 (Estimated); Primary Completion 2018-02-19 (Estimated); Study Completion 2018-08-19 (Estimated)

PRIMARY OUTCOMES:
sulcus bleeding index | baseline, change from baseline sulcus bleeding index at 4 weeks, change from baseline sulcus bleeding index at 8 weeks
  bleeding upon probing of gingival sulcus from the most severe periodontitis tooth

CONTACTS AND LOCATIONS:
Overall Officials: Nis Okuma, DDS, MD, M.Sc (Oral Medicine), Principal Investigator — Mahidol University
Locations (1):
- Burapha University Hospital, Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Undecided